CLINICAL TRIAL: NCT03342066
Title: Reproducibility of Interactive Cariogram Software Versus Manual Caries Risk Assessment Form on Clinician Decision: Observational Study
Brief Title: Reproducibility of Interactive Cariogram Software Versus Manual Caries Risk Assessment Form
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Gamal ashour, Dentist, Cairo University
Other Study IDs: gsda.1986
Record Dates: First submitted 2017-11-06; First posted 2017-11-14 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — bacteria isolated from saliva
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A: Cariogram
  Interventions: Diagnostic Test: reproducability of caries risk assessment
- B: CAMBRA
  Interventions: Diagnostic Test: reproducability of caries risk assessment

INTERVENTIONS:
Diagnostic Test: reproducability of caries risk assessment — reproducability of caries risk assessment CAMBRA verses cariogram

SUMMARY:
Reproducibility of Interactive Cariogram Software versus Manual Caries Risk Assessment Form on Clinician Decision: observational study

DETAILED DESCRIPTION:
A main factor for planning any preventive program is to accurately assess a person's risk of developing a caries. Dental caries is a multifactorial disease and is affected by several factors, such as the patient's general health and diet, the amount and type of bacteria present in the oral cavity, salivary factors and exposure to fluoride.

Thus, caries risk assessment approaches should take into account risk implications from various factors that influence carious activity Many caries risk assessment models had been developed to assess the caries for certain individual, this study will be carried out to measure the reproducibility between CAMBRA and cariogram model to evaluate if one of them is enough to be used as they give the same result or not

ELIGIBILITY:
Inclusion Criteria:

* Patients should be in range of 18-40 years old. Patient should have good periodontal health

Exclusion Criteria:

* Patient below 18 years and above 40 years old Patient with periodontally affected teeth and mobility. Patient with multiple extraction

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: patients of both sex ,age from 18-40 with different oral hygiene and different dental condition but with good periodontal condition and no multiple extraction
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-02-10 (Actual); Study Completion 2019-02-10 (Actual)

PRIMARY OUTCOMES:
Reproducability "degree of matching between cariogram and cambra | one day
  reproducability of cariogram and cambra

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed farid, prof.Dr, Study Director — Professor, Conservative Dentistry Department, Faculty of dentistry, Cairo University, Egypt.
Locations (1):
- Cairo Univeristy, Cairo, Manial, Egypt